CLINICAL TRIAL: NCT01336192
Title: Maintenance Gemcitabine or Best Supportive Care for the Chinese Advanced NSCLC Patients Without Progression Disease After Given Four Cycles of the Induction Chemotherapy With Gemcitabine Plus Cisplatin
Brief Title: Maintenance Gemcitabine in the Chinese Advanced Lung Cancer
Acronym: MAGICAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Di Zheng/MD, Shanghai Pulmonary Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHPH-11ZL113
Record Dates: First submitted 2011-04-07; First posted 2011-04-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Advanced NSCLC; Maintenance therapy; Gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best supportive care (No Intervention): Best supportive care
- Maintenance gemcitabine (Experimental): Maintenance therapy of gemcitabine alone
  Interventions: Drug: Gemcitabine; Drug: Best supportive care

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1250mg/m^2 Day 1 and 8, 28 days per cycle until PD
  Arms: Maintenance gemcitabine
Drug: Best supportive care — Best supportive care
  Arms: Maintenance gemcitabine

SUMMARY:
Lung cancer, the most common cancer worldwide, remains the leading cause of cancer death. Approximately two-thirds of all patients with newly diagnosed non-small-cell lung cancer (NSCLC) present with advanced stage that palliative chemotherapy is the only appropriate measure. The standard treatment for this patient population consists of third generation platinum-based doublet regimen for no more than 6 cycles followed by watch and wait until disease progression (PD) before the administration of second-line and third-line systemic anticancer therapeutic agents. Patients who go on to receive second-line therapy represent a selected subgroup with an improved overall prognosis.

Switch maintenance therapy with pemetrexed or erlotinib in patients with advanced NSCLC without PD after first-line chemotherapy has been confirmed to improve progression free survival (PFS) and overall survival (OS) significantly compared with placebo in two large randomized controlled studies. However, continuation gemcitabine maintenance therapy in this setting yields conflicting results in the west, i.e.showing a prolongation of PFS without OS improvement. Thus, we investigate the efficacy and safety of continuation of gemcitabine maintenance therapy for patients with metastatic NSCLC with ECOG performance status of 0-1 and without PD after four cycles of first-line chemotherapy with gemcitabine and cisplatin in China.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmed diagnosis of Stage IV NSCLC according to 2009 the seventh edition of TNM staging of lung tumors.
* No disease progression after four cycles of first-line chemotherapy with gemcitabine plus cisplatin (running period) within one month before the enrollment.
* Brain metastases are permitted if treated with full course of whole brain radiotherapy without the presence of symptomatic central nervous system metastases.
* ECOG score 0-1

Exclusion Criteria:

* First-line chemotherapy other than combination treatment of gemcitabine plus cisplatin
* Other therapy including targeted therapy, immunotherapy and prior radiotherapy for the treatment of the primary tumor prior to enrollment.
* Active infection
* Inadequate liver and renal function.
* Serious concomitant systemic disorder incompatible with the study.
* Second primary malignancy (except in situ carcinoma of the cervix, adequately treated basal cell carcinoma of the skin, T1 vocal cord cancer in remission, or prior malignancy treated more than 5 years prior enrollment without recurrence)
* Presence of the pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  From the start of maintenance therapy or Best Suppotive Care(BSC) until the date of documented progressive disease or death from any cause

SECONDARY OUTCOMES:
Overall Survival | 18 months
  From the start of maintenance therapy or BSC until the date of documented death from any cause
Response Rate | approximately 4 weeks
  From the start of maintenance therapy or BSC until the date of documented progressive disease
Time to The Progression | 18 months
  From the start of maintenance therapy or BSC until the date of documented progressive disease
Health Related Quality of Life | Approximately 4 weeks
  From the start of maintenance therapy or BSC until the date of documented progressive disease or the termination of study
Number of Participants with treatment-related grade III/IV adverse events | 6 months
  frequency and severity of adverse events and laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Di Zheng, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Wen Gao, MD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China; Jianfang Xu, MD, Study Director — Shanghai Pulmonary Hosptial; Li Wang, MD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China; Meijun Lv, MD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China; Jian Ni, MD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China; Jie Zhang, MD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China; Bing Lu, MD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China; Ying Xu, MD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital Medical Oncology Department, Shanghai, Shanghai Municipality, China